CLINICAL TRIAL: NCT03414203
Title: Comparison Between Stimulation Transcranial Protocols With Continuous Current in the Chronic Migraine: Clinical Trial, Triple-blind, Placebo-controlled
Brief Title: Comparison Between Transcranial Stimulation Protocols With Continuous Current in the Chronic Migraine
Acronym: NEUROMIG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Paraíba (Other)
Responsible Party: Principal Investigator, Renata Emanuela Lyra de Brito Aranha, researcher, Federal University of Paraíba
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NEUROMIG
Record Dates: First submitted 2018-01-10; First posted 2018-01-29 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Chronic Migraine
Keywords: Transcranial Direct Current Stimulation; Migraine Disorders; Cognitive Symptoms
MeSH Terms: conditions — Migraine Disorders; Neurobehavioral Manifestations | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: The patients will be randomized into 1 of 3 groups:
  group A: active tDCS for 15 minutes, group B: active tDCS for 15 minutes, with an interval of 20 minutes and group C: more 15 minutes os stimulation, sham tDCS for 15 minutes.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- active tDCS (Active Comparator): Active tDCS for 15 minutes for 10 days over 2 weeks. Intensity: 2 milliampere. Placement: anode - left DLPFC; cathode - right supraorbital region
  Interventions: Other: tDCS
- active tDCS with interval (Experimental): Active tDCS for 15 minutes, interval of 20 minutes and more 15 minutes for 10 days over 2 weeks. Intensity: 2 milliampere. Placement: anode - left DLPFC; cathode - right supraorbital region
  Interventions: Other: tDCS
- sham tDCS (Sham Comparator): Sham tDCS for 15 minutes for 10 days over 2 weeks. The stimulation is non-active. Placement: anode - left DLPFC; cathode - right supraorbital region
  Interventions: Other: tDCS

INTERVENTIONS:
Other: tDCS — Transcranial Current Stimulation equipment consists of an ammeter (measured with current intensity), a potentiometer (voltage controller between the electrodes), a generator (two 9-volt batteries) and two electrodes (anode and cathode). The direct low-amplitude currents released by the electrodes reach the cortex and modify the neuronal potentials.

SUMMARY:
This study aims to compare the effects of transcranial direct current stimulation on the clinical and cognitive function in patients with chronic migraine.

DETAILED DESCRIPTION:
The patients will be randomized into 1 of 3 groups: active tDCS for 15 minutes, active tDCS for 15 minutes, with an interval of 20 minutes and more 15 minutes os stimulation, sham tDCS for 15 minutes. The tDCS will be applied for 10 days over 2 weeks.

ELIGIBILITY:
Inclusion Criteria:

* females
* clinical diagnosis of chronic migraine according to the International Classification of Headaches Disorders (ICHD-3 beta).

Exclusion Criteria:

* headache attributable to some pathological condition, associated neurologic or neuropsychiatric disease
* use of central nervous system modulating drugs
* pregnancy
* metallic head implants
* use of a cardiac pacemaker

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2017-08-14 (Actual); Primary Completion 2018-02-05 (Actual); Study Completion 2018-02-16 (Actual)

PRIMARY OUTCOMES:
Migraine Disability Assessment - MIDAS | "before treatment", "after treatment - up to 2 weeks " and "up to 1 month after the last day of treatment"
  Change in perform activities of daily living associate to migraine assessed on the Migraine Disability Assessment - MIDAS.

SECONDARY OUTCOMES:
Headache Impact Test - HIT-6 | "before treatment", "after treatment - up to 2 weeks " and "up to 1 month after the last day of treatment"
  Change in quality of life associate to migraine assessed on the Headache Impact Test-6 (HIT-6)
Wechsler Intelligence Scale Letters | "before treatment", "after treatment - up to 2 weeks " and "up to 1 month after the last day of treatment"
  Change in cognitive ability assessed on the Wechsler Adult Intelligence Scale Letters
Wechsler Intelligence Scale Numbers Test | "before treatment", "after treatment - up to 2 weeks " and "up to 1 month after the last day of treatment"
  Change in cognitive ability assessed on the Wechsler Adult Intelligence Scale Numbers Test
Hayling's Test Hayling's Test | "before treatment", "after treatment - up to 2 weeks " and "up to 1 month after the last day of treatment"
  Change in operational memory assessed on the Hayling's Test Evaluate operational memory
Trail Making Test part B | "before treatment", "after treatment - up to 2 weeks " and "up to 1 month after the last day of treatment"
  Change in executive functions assessed on the Trail Making Test part B
Salthouse Visual Patterns and Lyrics | "before treatment", "after treatment - up to 2 weeks " and "up to 1 month after the last day of treatment"
  Change in visual processing speed assessed on the Salthouse Visual Patterns and Lyrics
Nine Hole Peg Test | "before treatment", "after treatment - up to 2 weeks " and "up to 1 month after the last day of treatment"
  Change in the motor processing speed assessed on the Nine Hole Peg Test
Paced Auditory Serial Addition Task | "before treatment", "after treatment - up to 2 weeks " and "up to 1 month after the last day of treatment"
  Change in selective attention assessed on the Paced Auditory Serial Addition Task
Concentrated Attention Test | "before treatment", "after treatment - up to 2 weeks " and "up to 1 month after the last day of treatment"
  Change in selective attention assessed on the Concentrated Attention Test
Visual Attention Test (Attention Matrices) | "before treatment", "after treatment - up to 2 weeks " and "up to 1 month after the last day of treatment"
  Change in selective attention assessed on the Visual Attention Test (Attention Matrices)
Montreal Cognitive Assessment | "before treatment", "after treatment - up to 2 weeks " and "up to 1 month after the last day of treatment"
  Change in cognition assessed on the Montreal Cognitive Assessment
Side Effects Questionnaire | "every day for up to 2 weeks"
  adverse effects assessment

CONTACTS AND LOCATIONS:
Overall Officials: Renata Aranha, Principal Investigator — Federal University of Paraiba
Locations (1):
- Federal University of Paraiba, João Pessoa, Paraíba, Brazil